CLINICAL TRIAL: NCT06733792
Title: Efficacy of a Digitalized Selective Prevention Program (App - "CANQUIT") to Reduce and/or Quit Cannabis Use
Brief Title: A Mobile App to Reduce and/or Quit Cannabis Use
Acronym: CANQUIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alba González-Roz, PhD (Other)
Collaborators: Delegación del Gobierno para el Plan Nacional sobre Drogas (Unknown)
Responsible Party: Sponsor-Investigator, Alba González-Roz, PhD, PhD, Associate Professor, University of Oviedo
Organization: University of Oviedo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-23-PNSD-1; 2022I002 (Other Grant/Funding Number: Government Delegation for the National Plan on Drugs)
Record Dates: First submitted 2024-12-06; First posted 2024-12-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cannabis Dependence
Keywords: Cannabis; App-based intervention; Young adults; Selective prevention; CBT; Contingency Management
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App-assisted CBT-based intervention (Experimental): Participants have access to a 4-week digitalized CBT-based intervention. Participants will have access to seven weekly modules. Modules include cannabis-related psychoeducation (i.e., benefits concerning cannabis use reduction/quitting, short- and long-term consequences, myths), training in emotional regulation strategies, stimulus control (i.e., alternatives to cannabis use), behavioral activation strategies and relapse prevention (i.e., training in assertiveness skills and problem-solving abilities).
  Interventions: Behavioral: CBT-based intervention
- App-assisted self-help guide (Active Comparator): Participants receive a self-help guide based on psychoeducation on cannabis use and its physical/mental health effects.
  Interventions: Behavioral: Self-help guide

INTERVENTIONS:
Behavioral: CBT-based intervention — * 1st week: Daily self-report on cannabis and tobacco use, myths regarding cannabis use and its health consequences, motives for cannabis use reduction/quitting, psychoeducation concerning withdrawal symptomatology, therapist's recommendation (progressive reduction of cannabis use).
  * 2nd week: Daily self-report on cannabis and tobacco use, myths regarding cannabis use and its health and behavioral consequences, identification of triggers, alternatives to cannabis use, therapist's recommendation (progressive reduction of cannabis use).
  * 3rd week: Daily self-report on cannabis and tobacco use benefits from quitting cannabis, behavioral activation, diaphragmatic breathing, training in social abilities, strategies to prevent smoking, therapist's recommendation (progressive reduction of cannabis use).
  * 4th week: Daily self-report on cannabis and tobacco use (i.e., nº of joints/cigarettes), high-risk situations for relapse, lapse vs. relapse, coping strategies, relapse prevention plan.
  Arms: App-assisted CBT-based intervention
Behavioral: Self-help guide — Psychoeducation on cannabis.
  Arms: App-assisted self-help guide

SUMMARY:
This study aims to develop an App-based intervention (CANQUIT) aimed at regular cannabis users. The efficacy of this intervention will be evaluated in the short-term (1-month follow-up) and long-term (3- and 6-months follow-ups) using a sample of 120 participants. Participants will be randomly assigned to the experimental arm (App-assisted CBT-based intervention) or the control (App-assisted self-help guide). The study will also estimate the economic impact of the intervention by considering the benefit-cost ratio (BCR) and net benefit (in €) associated with the total cost of the program. The goal is to provide evidence that can inform policy decisions regarding cannabis use and minimize the negative consequences on the physical and mental health of young adults in Spain. This study aims to offer a cost-effective prevention strategy that minimize the negative consequences on the physical and mental health of young adults in Spain.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy and cost-effectiveness in the short (1-month) and long-term (3 and 6 months) of a digitalized intervention (CANQUIT) to reduce and/or quit cannabis among young Spanish adults.

CANQUIT is a 4-week digitalized CBT-based intervention aimed at reducing or ceasing cannabis use among regular cannabis users (at least 1 occasion of cannabis use in the previous month). It is specifically tailored to young adults (18-30 years old). CANQUIT will be available to download both on Apple Store (iOS) and Play Store (Android). Upon completion of the baseline assessment, participants will be randomly assigned 2:1 to either an experimental arm (60 participants: App-assisted CBT-based intervention) or control (60 participants: App-assisted self-help guide). Participants in the experimental arm will be exposed to seven weekly modules, which include: 1) psychoeducation regarding the benefits of ceasing cannabis use, its short and long-term effects and myths associated with its consumption, 2) training in emotion regulation strategies, stimulus control (i.e., alternatives to cannabis use), 3) behavioral activation strategies, and 4) relapse prevention (i.e., assertiveness and problem-solving abilities). Participants will also register daily consumption of cannabis (number of joints) and receive weekly recommendations regarding cannabis use reduction. To ensure adherence to treatment, CANQUIT includes gamification via direct contact with a mental health professional and social interaction with others (through an online chat).

Alternatively, participants allocated to the control group will receive a self-help guide with information based on the contents of the App. This guide will be also available through the App. As in the experimental arm, participants in the control group will also complete 1-month, 3-months and 6-months follow-ups through the App.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 30 years old.
* At least one occasion of cannabis use in the last month.
* Access to smartphones (iOS or Android).
* Access to Internet.

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cannabis abstinence | 7-day point prevalence abstinence (PP) at 4-week follow-up (FU), 3-months follow-up (FU), 6-months follow-up (FU)
  * Self-reported point prevalence cannabis abstinence
  * Continuous self-reported cannabis abstinence
Cannabis reduction | 4 weeks follow-up (FU), 3 months follow-up (FU), 6 months follow-up (FU)
  * Self-reported reduction in quantity of cannabis used on a weekly basis (daily joints, number of hashish/marijuana joints, grams)
  * Decreases in self-reported past-month frequency of cannabis use (i.e., once, less than one per week, once/twice per week, 3-4 times a week, 5-6 times a week, every day).
Acceptability | 4-week follow-up (FU)
  Client Satisfaction Questionnaire-8 (CSQ-8). The CSQ-8 is an 8-item questionnaire that evaluates the level of satisfaction with the treatment received by the participants. Scores range between 8-32, with higher scores indicating higher levels of satisfaction.

SECONDARY OUTCOMES:
Changes in legal and illegal substance use | 4 weeks follow-up (FU), 3 months follow-up (FU), 6 months follow-up (FU),
  Self-reported past-month legal and illegal substance use (alcohol, tobacco, cocaine, heroine, amphetamine, ecstasies, hallucinogens, prescription drugs).
Changes in cannabis-related problems | 4-week follow-up (FU), 3-months follow-up (FU), 6-months follow-up (FU)
  Pre to post-intervention changes in cannabis problems as measured by the Cannabis Use Disorder Identification Test-Revised (CUDIT-R). The CUDIT-R is an 8-item screening test for measuring cannabis-related problems. Scores of 8 or more are indicative of hazardous cannabis use. Meanwhile, scores of 12 or more indicate the participant may present a cannabis use disorder.
Improvement in risk of emotional disorders | Changes in 4-week follow-up (FU), 6-months follow-up (FU)
  Reductions in the severity of symptoms of depression, anxiety, somatization as measured by the Brief Symptoms Inventory-18 (BSI-18). The BSI-18 is an 18-item assessment screening of psychological distress (somatic, anxious and depressive symptomatology). Scores range between 0-72, with higher values indicating higher risk of depression, anxiety and somatization.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Faculty of Psychology, University of Oviedo, Oviedo, Principality of Asturias
  - University of Oviedo, Oviedo, Principality of Asturias

REFERENCES:
- [Background] Derogatis, L.R. (2001). BSI 18, Brief Symptom Inventory 18: Administration, scoring and Procedure Manual. Pearson.
- [Background] Adamson SJ, Kay-Lambkin FJ, Baker AL, Lewin TJ, Thornton L, Kelly BJ, Sellman JD. An improved brief measure of cannabis misuse: the Cannabis Use Disorders Identification Test-Revised (CUDIT-R). Drug Alcohol Depend. 2010 Jul 1;110(1-2):137-43. doi: 10.1016/j.drugalcdep.2010.02.017. Epub 2010 Mar 26. PMID 20347232
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963